CLINICAL TRIAL: NCT00901641
Title: Computer-Based Cognitive Training and Sleep Quality in Older Adult Insomniacs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Max Stern Academic College Of Emek Yezreel (Other)
Responsible Party: Haimov Iris, Ph.D.,associate professor, The Max Stern Academic College Of Emek Yezreel
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: emek123-08
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Insomnia
Keywords: cognitive training; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive training (Experimental): CogniFit Personal Coach® computer cognitive training program. The program provides individually tailored cognitive training based on the results of a baseline evaluation (the Neuropsychological Examination - CogniFit Personal Coach®). The program assigns scores to 17 cognitive abilities that are subsequently trained by means of 21 different tasks.
  Interventions: Device: CogniFit Personal Coach®

INTERVENTIONS:
Device: CogniFit Personal Coach® — The program provides individually tailored cognitive training based on the results of a baseline evaluation (the Neuropsychological Examination - CogniFit Personal Coach®).7 The program assigns scores to 17 cognitive abilities that are subsequently trained by means of 21 different tasks.

SUMMARY:
The purpose of this study is to investigate the effect of computerized, home-based cognitive training on sleep quality of older adults with insomnia.

DETAILED DESCRIPTION:
Participants in the cognitive training group train in a computer-based cognitive training program over a period of 12 weeks. An active control group train in a program involving tasks that do not engage high-level cognitive functioning over the same period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic insomnia
* able to use a home personal computer
* have healthy dominant hand functioning
* Hebrew speakers

Exclusion Criteria:

* have any significant visual or hearing impairment
* have any significant medical, neurological or psychiatric illness that might bring about cognitive change
* have sleep disorders other than insomnia
* have any significant medical disease (including cancer, diabetes, liver, kidney, heart or lung disease)
* alcoholism or other drug abuse
* taking any medication known to affect central nervous system functioning other than sleeping pills
* historical evidence suggesting significant psychiatric conditions such as depression, psychosis or neurologic disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-05; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
sleep measures | 3-6 months

SECONDARY OUTCOMES:
Cognitive performance | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Iris Haimov, Ph.D., Principal Investigator — The Max Stern Academic College Of Emek Yezreel
Locations (1):
- The Max Stern Academic College of Emek Yezreel, Emek Yezreel, Israel

REFERENCES:
- [Background] Haimov I, Hanuka E, Horowitz Y. Chronic insomnia and cognitive functioning among older adults. Behav Sleep Med. 2008;6(1):32-54. doi: 10.1080/15402000701796080. PMID 18412036
- [Derived] Haimov I, Shatil E. Cognitive training improves sleep quality and cognitive function among older adults with insomnia. PLoS One. 2013;8(4):e61390. doi: 10.1371/journal.pone.0061390. Epub 2013 Apr 5. PMID 23577218